CLINICAL TRIAL: NCT04380831
Title: Pilot Study of Total Body Irradiation Using Intensity Modulated Radiation Therapy (IMRT) and Cyclophosphamide Conditioning Regimen Prior to Autologous Hematopoietic Cell Transplantation in Patients With Severe Systemic Sclerosis
Brief Title: TBI Using IMRT and Cyclophosphamide Prior to Stem Cell Transplant for the Treatment of Severe Systemic Sclerosis
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20006; NCI-2020-02744 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20006 (Other: City of Hope Medical Center)
Record Dates: First submitted 2020-04-30; First posted 2020-05-08 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Systemic Scleroderma
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Stem Cell Transplantation; Cyclophosphamide; Radiotherapy, Intensity-Modulated; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (TBI using IMRT, cyclophosphamide, HSCT) (Experimental): Patients undergo TBI using IMRT BID on days -5 and -4 in the absence of disease progression or disease progression. Patients then receive cyclophosphamide on days -3 and -2 and undergo HSCT on day 0 in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Cyclophosphamide; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Total-Body Irradiation

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo HSCT
  Other Names: Allogeneic Hematopoietic Cell Transplantation; allogeneic stem cell transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
Drug: Cyclophosphamide — Undergo HSCT
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Radiation: Intensity-Modulated Radiation Therapy — Undergo TBI using IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Procedure: Total-Body Irradiation — Undergo TBI using IMRT
  Other Names: TBI; Total Body Irradiation; Whole Body Irradiation; Whole-Body Irradiation

SUMMARY:
This early phase I trial studies the side effects and feasibility of total body irradiation using intensity modulation radiation therapy (IMRT) when given in combination with cyclophosphamide prior to stem cell transplant to treat severe systemic sclerosis. IMRT delivers total body radiation therapy more precisely and may reduce radiation exposure to sensitive normal organs. Giving chemotherapy, such as cyclophosphamide, and total body irradiation before a donor stem cell transplant helps kill cancer cells in the body and helps make room in the bone marrow for new blood-forming cells (stem cells) to grow. Giving IMRT and cyclophosphamide prior to stem cell transplant may work better in treating severe systemic sclerosis and reduce radiation doses to lung and kidneys compared to cyclophosphamide alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility of using IMRT to deliver total body irradiation (TBI) to 800 cGy while keeping mean lung and kidney doses to 200 cGy.

II. To assess the safety/feasibility of total body irradiation using IMRT (IMRT TBI) in systemic sclerosis patients undergoing autologous hematopoietic stem cell transplantation.

SECONDARY OBJECTIVES:

I. To evaluate dose homogeneity and dose sparing to lung and kidneys. II. To evaluate transplant-related mortality at 30 days and 100 days post IMRT TBI.

OUTLINE:

Patients undergo TBI using IMRT twice daily (BID) on days -5 and -4 in the absence of disease progression or disease progression. Patients then receive cyclophosphamide on days -3 and -2 and undergo HSCT on day 0 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up on days 30 and 100.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky performance status (KPS) >= 70
* Systemic sclerosis patients evaluated within 30 days of start of conditioning regimen who would be candidates for TBI-cyclophosphamide (Cy) per City of Hope (COH) guidelines and standard operating procedures (SOP) for autologous hematopoietic cell transplant
* Patients must be suitable for TBI conditioning regimens as part of transplant per radiation the referring hematologist
* Patients must have adequate organ function for HCT as determined by the hematologist
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation
* All subjects must have the ability to understand the treatment and the willingness to sign a written informed consent

Exclusion Criteria:

* Patients should not have any uncontrolled illness including ongoing or active infection
* Prior history of radiation therapy must be presented to study principal investigator (PI) for eligibility determination
* Pregnant women are excluded from this study because total body irradiation is an agent with the potential for teratogenic or abortifacient effects
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-02-24 (Actual); Primary Completion 2026-12-22 (Estimated); Study Completion 2026-12-22 (Estimated)

PRIMARY OUTCOMES:
Mean lung dose | Up to day 100
  The study will be deemed feasible if >= 80% of patients complete the intensity modulation radiation therapy (IMRT) to the total dose of 800 cGy, mean lung and kidney doses are limited to 200 cGy or less.
Mean kidney dose | Up to day 100
  The study will be deemed feasible if >= 80% of patients complete the IMRT to the total dose of 800 cGy, mean lung and kidney doses are limited to 200 cGy or less.

SECONDARY OUTCOMES:
Dose homogeneity for lungs, kidneys, and total body | Up to day 100
  "Dose homogeneity for lung, kidney and total body will use the DVH (dose volume histograms) generated by the treatment plan for each of these regions. The goal is to keep the lung and kidney dose homogeneity to with +/- 15% of the mean dose to that organ. The goal is to keep total body dose homogeneity to within +/- 15% of the prescribed total body dose of 8 Gy."
Transplant-related mortality | Day 30 and day 100
  Measured by comparing the transplant-related mortality rates on day 30 compared to day 100.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Y Wong, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States